CLINICAL TRIAL: NCT01374477
Title: Hypertensive Disorders of Pregnancy in Adolescence and the Primipaternity Concept. Cases and Control Trial
Brief Title: Hypertensive Disorders of Pregnancy in Adolescence and Primipaternity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., MD, Saint Thomas Hospital, Panama
Other Study IDs: MHST2011-05
Record Dates: First submitted 2011-06-14; First posted 2011-06-16 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2015-01

CONDITIONS: Preeclampsia
Keywords: Preeclampsia in Adolescence; Adolescent; Primipaternity
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Adolescent with preeclampsia: Patients < 19 years old who delivered in our institution (vaginal birth or cesarean) that developed a hypertensive disorder of pregnancy.
- Normal adolescent: Patients < 19 years old who delivered in our institution (vaginal birth or cesarean) without developing a hypertensive disorder of pregnancy.

SUMMARY:
Hypertensive disorders of pregnancy are one of the most frequent complications of pregnancy, being a serious health problem around the world.

Previous studies have suggested that there is an association between a short period of exposure to paternal sperm of a new sexual partner and the development of an immunological reaction that could trigger a hypertensive disorder of pregnancy. For this reason we want to study the relationship between the primipaternity concept (exposure to male antigens present in semen over a short period of time previous to the pregnancy) and the development of preeclampsia in adolescents.

ELIGIBILITY:
Inclusion Criteria:

* 19 year old or less
* Pregnancy > 24 weeks at the moment of delivery

Exclusion Criteria:

* 20 years old or more.
* Pregnancy < 24 weeks at the moment of delivery

Max Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients < 19 years old who delivered in our institution.
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2012-06; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Presence of a primipaternity factor | Two months
  The presence of primipaternity factor. They include:
  1. Sexual Cohabitation (timeframe between first sexual intercourse and pregnancy < 4 months)without the use of a barrier contraceptive.
  2. Oral sex with ejaculation (previous to pregnancy < 4 months).

SECONDARY OUTCOMES:
Maternal complications | Two months
  Presence of a complication related to preeclampsia: abruptio placenta, HELLP syndrome, eclampsia.

CONTACTS AND LOCATIONS:
Overall Officials: Osvaldo Reyes, MD, Principal Investigator — Saint Thomas Hospital, Panama
Locations (1):
- Saint Thomas Hospital, Panama City, Provincia de Panamá, Panama